CLINICAL TRIAL: NCT05924217
Title: Gynecology Beyond Gender: Exploration and Identification of Potential Obstacles and Levers in France for Cervical Cancer Screening in Transgender Men, by Conducting an Opinion Survey in a Specific Population
Brief Title: Gynecology Beyond Gender: Cervical Cancer Screening in Transgender Men in France
Acronym: GYDECAT
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2023/thése/IJ-01
Record Dates: First submitted 2023-06-12; First posted 2023-06-29 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer; Transgender Persons; Health Services for Transgender Persons
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey questionnaire — This survey aims to explore the perception that transgender men have of cervical cancer screening and to identify the challenges they face, the obstacles and the levers to access this prevention program.

SUMMARY:
In France, cervical cancer screening is the subject of a national screening programme organized for all asymptomatic individuals aged 25 to 65 years with a cervix. The latter contributes greatly to the prevention and early treatment of this disease, whose public health challenge is recognized worldwide.

One of the objectives of this programme is to reduce inequalities in access. Transgender men, i.e. individuals assigned to the female gender at birth but identifying with the male gender, are concerned by this screening as long as they still have a cervix, according to the same modalities as for cisgender women.

However, they are often excluded from health care, including organized screening programs. Gender change in civil status is one of the obstacles.

The provision of gynaecological care is sometimes inadequate. The lack of knowledge of health professionals and the problems of discrimination that transgender people may face reduce the chances of having equitable access.

This survey aims to explore the perception that transgender men have of cervical cancer screening and to identify the challenges they face, the obstacles and the levers to access this prevention program.

ELIGIBILITY:
Inclusion Criteria:

* transgender male (assigned female at birth but identifying as male)
* aged 25 to 65 years
* Having retained her cervix
* Having had sex before.

Exclusion Criteria:

* Under 25 and over 65
* Not having retained his cervix
* History of cancerous lesion of the cervix

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transgender men, i.e. individuals assigned the female gender at birth but identifying with the male gender, who retained the cervix
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of transgender men who have ever been screened for cervical cancer in their lifetime | At study entry, basline (no follow-up)
  answer yes to the question "Have you ever been screened for cervical cancer in your lifetime?"

SECONDARY OUTCOMES:
prevalence of transgender men who feel concerned about cervical cancer screening | At study entry, basline (no follow-up)
  answer yes to the question "Do you feel personally involved in cervical cancer screening?"

CONTACTS AND LOCATIONS:
Overall Officials: ingrid JULIER, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France